CLINICAL TRIAL: NCT05910047
Title: The Effects of Six-week Hydrogen Plus Pyrroloquinoline Quinone (PQQ) Intake on Mitochondrial Biomarkers, Brain Metabolism and Cognition in the Elderly With Mild Cognitive Impairment
Brief Title: Supplemental Hydrogen Plus PQQ for Mitochondrial Biomarkers and Brain Function in Elderly With Mild Cognitive Impairment
Acronym: CALERIE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Novi Sad, Faculty of Sport and Physical Education (Other)
Responsible Party: Principal Investigator, Sergej Ostojic, Professor, University of Novi Sad, Faculty of Sport and Physical Education
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: A13-CH-2023
Record Dates: First submitted 2023-06-08; First posted 2023-06-18 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Age-associated Memory Impairment
Keywords: MITOCHONDRIAL BIOMARKERS; BRAIN METABOLISM; COGNITION
MeSH Terms: interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supplement (Experimental): One tablet of supplement before breakfast and dinner
  Interventions: Dietary Supplement: Supplement
- Placebo (Placebo Comparator): One tablet of inert compound before breakfast and dinner
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Supplement — Dietary supplement containing molecular hydrogen and pyrroloquinoline quinone
  Arms: Supplement
Dietary Supplement: Placebo — Inert substance
  Arms: Placebo

SUMMARY:
The goal of this randomized controlled double-blind parallel-group interventional trial is to evaluate the effects of dietary supplementation with molecular hydrogen and pyrroloquinoline quinone in elderly. The main questions it aims to answer are: (1) whether the supplementation affects biomarkers of mitochondrial function in serum, and (2) whether the supplementation affects cognition and brain metabolism. The participants will be subjected to take the dietary supplement during 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age > 65 years
* MMSE scores ranged from 23-27
* Informed consent signed

Exclusion Criteria:

* Take part in exercise on a regular basis
* Severe chronic disease and acute injuries
* History of dietary supplement use during the past 4weeks
* No consent to randomization
* Participation in other studies

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Fibroblast growth factor 21 | Change from baseline serum fibroblast growth factor 21 at 6 weeks
  Level of fibroblast growth factor 21 in serum

SECONDARY OUTCOMES:
Peroxisome proliferator-activated receptor gamma coactivator 1-alpha | Change from baseline serum peroxisome proliferator-activated receptor gamma coactivator 1-alpha at 6 weeks
  Level of peroxisome proliferator-activated receptor gamma coactivator 1-alpha 21 in serum
Brain-derived neurotrophic factor | Change from baseline serum brain-derived neurotrophic factor at 6 weeks
  Level of brain-derived neurotrophic factor in serum
Irisin | Change from baseline serum irisin at 6 weeks
  Level of irisin in serum
General cognition | Change from baseline MMSE score at 6 weeks
  Mini-MentalStateExamination (MMSE) score
Brain creatine | Change from baseline brain creatine at 6 weeks
  MRS spectra for brain creatine
Brain oxygenation | Change from baseline brain oxygenation at 6 weeks
  Near-infrared spectroscopy for prefrontal oxygen saturation

CONTACTS AND LOCATIONS:
Locations (1):
- FSPE Applied Bioenergetics Lab, Novi Sad, Vojvodina, Serbia

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in age-related mild cognitive impairment. Data will be coded, with no PHI included. Approval of the request and execution of all applicable agreements are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.

REFERENCES:
- [Background] Zanini D, Todorovic N, Korovljev D, Stajer V, Ostojic J, Purac J, Kojic D, Vukasinovic E, Djordjievski S, Sopic M, Guzonjic A, Ninic A, Erceg S, Ostojic SM. The effects of 6-month hydrogen-rich water intake on molecular and phenotypic biomarkers of aging in older adults aged 70 years and over: A randomized controlled pilot trial. Exp Gerontol. 2021 Nov;155:111574. doi: 10.1016/j.exger.2021.111574. Epub 2021 Oct 1. PMID 34601077
- [Background] Ostojic SM. Does drinking water rich in hydrogen gas revive brain hypometabolism in neurodegeneration by SCFAs upregulation? Eur J Clin Nutr. 2021 Jan;75(1):212-213. doi: 10.1038/s41430-020-0680-x. Epub 2020 Jul 6. No abstract available. PMID 32632247
- [Background] Korovljev D, Stajer V, Javorac D, Ostojic SM. Hydrogen inhalation positively affects cardiometabolic risk factors in men and women aged 65 years or older: a preliminary report. Eur Geriatr Med. 2018 Oct;9(5):729-730. doi: 10.1007/s41999-018-0087-6. Epub 2018 Jul 31. No abstract available. PMID 34654221
- [Background] Korovljev D, Trivic T, Drid P, Ostojic SM. Molecular hydrogen affects body composition, metabolic profiles, and mitochondrial function in middle-aged overweight women. Ir J Med Sci. 2018 Feb;187(1):85-89. doi: 10.1007/s11845-017-1638-4. Epub 2017 May 30. PMID 28560519
- [Background] Ostojic SM. Targeting molecular hydrogen to mitochondria: barriers and gateways. Pharmacol Res. 2015 Apr;94:51-3. doi: 10.1016/j.phrs.2015.02.004. Epub 2015 Feb 24. PMID 25720951